CLINICAL TRIAL: NCT03059576
Title: Circadian System Heritability Assessed in Free Living Conditions in a Twin Mediterranean Population
Brief Title: Circadian System Heritability Assessed in Free Living Conditions
Acronym: MTR
Status: Completed | Type: Observational
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, PROF. MARTA GARAULET AZA, Proffesor, Universidad de Murcia
Other Study IDs: 2017ES00002
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: Chronobiology; Circadian rhythms; Heritability; Twins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Chronobiological status of the subjects — Participation was completely voluntary and not remunerated. The subjects were organized into groups of 5 pairs, and were given an appointment at a university facility located in the city center, where informed consent was signed prior to the procedures indicated below. An informational letter was sent to pre-selected individuals. Later a phone call confirmed their availability.
  * Temperature rhythm was assessed continuously for 7 days using a temperature sensor and programmed to collect information every 10 min.
  * Body position and rest-activity rhythm were assessed over the same 7 days using a Acceleration Data Logger that record data every min and placed on the non-dominant arm by means of an elastic band, with its X axis parallel to the humerus bone.
  * Diet and sleep record were completed over the same week, their sleep schedules and their nutritional status.

SUMMARY:
The purpose of this investigation is to assess the role of the genetic and environmental factor on circadian system, in free living conditions by the use of a female twin population. With the results from this study, the investigators expect to advance in the understanding of the role of the endogenicity of the circadian system variables such as temperature, activity, sleep and timing of food intake as the main cause of the coincidence of the rhythms. However, the investigators expected that some parameters are still dependent on environment to a relevant extent and, hence, amenable to change through external interventions.

DETAILED DESCRIPTION:
Twin studies are a classic in the analysis of the relative contribution of genetic and environmental factors to behavior and other phenotypes. These models are most often used to separate genetic from environmental causes in the family resemblance methodology. These models based on twins have been previously carried out in chronobiology. In fact, during the years 1993 and 1994, Paul Linkowski et al., performed two relevant studies on the circadian system to analyze the relative contributions of hereditary and/or environmental factors of cortisol secretion and blood pressure, respectively, and concluded that genetic factors control some of the characteristics of cortisol and diastolic blood pressure circadian rhythmicity. The heritability of other circadian markers has also demonstrated such as morningness- eveningness (44%), sleep-related variables have also pointed to a relevant role of genetics with heritability estimates of sleep duration between 17% and 55%. However, to the investigators knowledge, the heritability of other relevant chronobiological markers, measured in free living conditions such as body temperature, actigraphy and sleep has not been studied.

These goals will be achieved through a specific approach:

* Observational (Aim 1): To study the potential effect of the genetic and environmental factor in the circadian system health in order to improve the chronobiological therapies in the clinical practice (n=106).

ELIGIBILITY:
IInclusion Criteria:

* Body Mass Index: >19 kg/m2
* Age: between 18 and 70 year of age
* Caucasian

Exclusion Criteria:

* Receiving treatment with thermogenic, lipogenic, or contraceptive drugs
* Diabetes mellitus, chronic renal failure, hepatic diseases, or cancer diagnosis
* Bulimia diagnosis, prone to binge eating
* Undergoing treatment with anxiolytic or antidepressant drugs

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All participants are voluntarily in the Murcia Twin Register in Spain. All participants are from the Spanish city of Murcia, located on the Southeast coast of the Mediterranean Sea.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Temperature record | Total of 1 week between Visit 1 and 2
  Measured using temperature sensor
Actigraphy record | Total of 1 week between Visit 1 and 2
  Measured using Pendant Acceleration Data Logger

SECONDARY OUTCOMES:
Light record | Total of 1 week between Visit 1 and 2
  Measured using Pendant Acceleration Data Logger
Sleep record | Total of 1 week between Visit 1 and 2
  Measured using Pendant Acceleration Data Logger

OTHER OUTCOMES:
Sleep Duration | Total of 1 week between Visit 1 and 2
  Sleep duration will be computed from self-reported
Total Energy Intake | Total of 1 week between Visit 1 and 2
  Total energy intake in kcal/day will be computed from 7-day 24-hr dietary recalls
Dietary Composition | Total of 1 week between Visit 1 and 2
  Macronutrient and micronutrient intake will be computed from 7-days of self-reported 24-hr dietary recalls
Dietary Intake Timing | Total of 1 week between Visit 1 and 2
  Food timing will be self-reported and averaged across 7-days of 24-hr dietary recalls
Chronotype | Total of 1 week between Visit 1 and 2
  Assessed using the Morningness-Eveningness Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Ramón, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez-Minguez J, Ordonana JR, Sanchez-Romera JF, Madrid JA, Garaulet M. Circadian system heritability as assessed by wrist temperature: a twin study. Chronobiol Int. 2015 Feb;32(1):71-80. doi: 10.3109/07420528.2014.955186. Epub 2014 Sep 10. PMID 25208247
- [Background] Lopez-Minguez J, Colodro-Conde L, Bandin C, Ordonana JR, Garaulet M, Madrid JA. Application of multiparametric procedures for assessing the heritability of circadian health. Chronobiol Int. 2016;33(2):234-44. doi: 10.3109/07420528.2015.1130051. Epub 2016 Jan 28. PMID 26817403
- [Derived] Lopez-Minguez J, Dashti HS, Madrid-Valero JJ, Madrid JA, Saxena R, Scheer FAJL, Ordonana JR, Garaulet M. Heritability of the timing of food intake. Clin Nutr. 2019 Apr;38(2):767-773. doi: 10.1016/j.clnu.2018.03.002. Epub 2018 Mar 12. PMID 29571565